CLINICAL TRIAL: NCT04199273
Title: Assessment of Human Diaphragm Strength by Magnetic and Electric Stimulation After Ultrasonography Phrenic Nerve Tracking : a Randomized, Cross Over, Physiologic Study in Critically Ill Patients Requiring Invasive Mechanical Ventilation
Brief Title: Assessment of Human Diaphragm Strength by Magnetic and Electric Stimulation After Ultrasonography Phrenic Nerve Tracking
Acronym: SONOSTIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: RECHMPL19_0202
Record Dates: First submitted 2019-12-09; First posted 2019-12-13 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Intensive Care Unit; Invasive Mechanical Ventilation
Keywords: Intensive Care Unit; Invasive Mechanical Ventilation; Diaphragm weakness assessment; Rehabilitation
MeSH Terms: interventions — Electric Stimulation

STUDY DESIGN:
Intervention Model Description: Each patient, serving as their own control, receives both types of phrenic nerve stimulation : magnetic stimulation and electric stimulation. The order is randomized. For avoid a carry-over effect (diaphragm potentiation), a wash-out period of 15 minutes will be respected between the two type of stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnetic stimulation and electric stimulation (Experimental): The patient receive first the magnetic stimulation with MagStim 200 tool. Then 15 min after he will receive the electric stimulation with the SonoStim tool : ultrasonography phrenic nerve tracking and targeted electric stimulation with a nerve stimulator usually used for neuromuscular transmission monitoring (TOFScan, Drager)
  Interventions: Procedure: Magnetic stimulation; Procedure: Electric stimulation
- Electric stimulation and magnetic stimulation (Experimental): The patient receive first electric stimulation with the SonoStim tool : ultrasonography phrenic nerve tracking and targeted electric stimulation with a nerve stimulator usually used for neuromuscular transmission monitoring (TOFScan, Drager). Then 15 min after he will receive the magnetic stimulation with MagStim 200 tool
  Interventions: Procedure: Magnetic stimulation; Procedure: Electric stimulation

INTERVENTIONS:
Procedure: Magnetic stimulation — Cervical bilateral phrenic nerve stimulation with the MagStim 200 tool.
Procedure: Electric stimulation — Cervical bilateral phrenic nerve stimulation after ultrasonography nerve tracking and targeted electric stimulation with a nerve stimulator usually used for neuromuscular transmission monitoring (TOFScan, Drager)

SUMMARY:
Development and validation of a new affordable and easy-to-use phrenic nerve stimulation tool for diaphragm strength assessment in intensive care unit

DETAILED DESCRIPTION:
In intensive care unit, various forms of sepsis, undernutrition, surgery, global inflammation, iatrogeny, and mechanical ventilation, contribute to the overall muscular involvement including the diaphragm.

Assessment of diaphragm dysfunction is a critical issue for patients under mechanical ventilation, providing prognosis information and leading to the best therapeutic choices.

Up to now, for sedated ventilated critical care patient, expensive magnetic phrenic nerve stimulation equipment is needed to evaluate diaphragm strength.

In this study, the investigators aim to develop an affordable easy-to-use phrenic nerve stimulation tool, with ultrasonography and a nerve stimulator usually used for neuromuscular transmission monitoring. Hypothesis is that phrenic pacing using this new method is equivalent to the Gold Standard.

ELIGIBILITY:
Inclusion Criteria:

* ICU patient with invasive mechanical ventilation
* Sedated patient with a Richmond Agitation-Sedation Scale of -4 or -5

Exclusion Criteria:

* Contraindication for magnetic stimulation (Pacemaker)
* Hemodynamic or respiratory instability : PaO2/FiO2 < 200 mmHg, noradrenaline > 0,3 µg/kg/min, dobutamine > 10 µg/kg/min
* Neuromuscular disease or recent use of neuromuscular blocking agents (2h30) with a TOF ratio below 4/4 95%.
* Refusal of study participation or to pursue the study by the patient, no consent
* Pregnancy or breastfeeding
* Absence of coverage by the French statutory healthcare insurance system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Tracheal pressure (Ptrach) during diaphragm pacing | During electric of magnetic phrenic nerve stimulation
  Negative pressure in the occluded breathing circuit, assessed with a manometer located just after the endotracheal tube, during diaphragm stimulation

SECONDARY OUTCOMES:
Behavioral Pain Scale (BPS) after stimulation | Immediately after phrenic nerve stimulation
  The BPS is a scale of pain for critical care patients, from 3 (no or minimal pain) to 12 points (maximum pain).
Distance in millimeter between anatomical and ultrasound phrenic nerve location | During ultrasonography phrenic nerve tracking
  Distance between classical anatomical landmarks of the phrenic nerve location (underneath the posterior border of the sternocleidomastoid muscle, at the level of the cricoid cartilage), and the phrenic nerve location with ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Samir Jaber, MD, PHD, Study Director — Montpellier University Hospital
Locations (1):
- Centre Hospitalier Universitaire Saint Eloi, Montpellier, Herault, France

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data will be made available upon a reasonable request
Supporting Information: Study Protocol
Time Frame: 12 months after the main publication
Access Criteria: Data are provided to qualified investigators free of charge. Required documents to request data include a summary of the research plan, request form, and institutional review board (IRB) review. Dataset will be shared after careful examination by the study board of investigators.

REFERENCES:
- [Derived] Capdevila M, De Jong A, Belafia F, Vonarb A, Carr J, Molinari N, Choquet O, Capdevila X, Jaber S. Ultrasound-guided Transcutaneous Phrenic Nerve Stimulation in Critically Ill Patients: A New Method to Evaluate Diaphragmatic Function. Anesthesiology. 2025 Mar 1;142(3):522-531. doi: 10.1097/ALN.0000000000005267. Epub 2024 Oct 21. PMID 39432817